CLINICAL TRIAL: NCT06831682
Title: Efficacy of Kinesiotaping During Rehabilitation Following Total Knee Replacement Surgery- a Prospective Randomised Controlled Trial
Brief Title: Efficacy of Kinesiotaping During Rehabilitation Following Total Knee Replacement Surgery
Acronym: KT-TKR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SRH Gesundheitszentrum Bad Herrenalb (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Study2024-BadHerrenalb-01
Record Dates: First submitted 2025-02-08; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Total Knee Replacement; Postoperative Recovery; Rehabilitation Outcome
Keywords: Kinesiotaping; Total Knee Replacement; Rehabilitation; knee joint Function; Pain Relief

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kinesiotaping group (Experimental): Patients in this group will receive Kinesiotaping (KT) in addition to standard rehabilitation following TKR surgery. KT will be applied using various techniques, including lymphatic, muscle, and ligament taping.
  Interventions: Device: Kinesiotaping (KT); Other: Standard Rehabilitation
- Control group (no KT) (Active Comparator): Patients in this group will receive standard rehabilitation following TKR surgery without the application of Kinesiotaping.
  Interventions: Other: Standard Rehabilitation

INTERVENTIONS:
Device: Kinesiotaping (KT) — Kinesiotaping will be applied using muscle, lymphatic, and ligament taping techniques to promote healing, reduce swelling, and improve muscle function following total knee replacement surgery.
  Other Names: K-Active Tape
  Arms: Kinesiotaping group
Other: Standard Rehabilitation — Patients will receive standard postoperative rehabilitation, including physiotherapy, gait training, and medical exercises, without the application of Kinesiotaping.

SUMMARY:
The aim of this study was to examine the efficacy of Kinesiotaping (KT) within postoperative rehabilitation after Total Knee Replacement (TKR) surgery by determining whether KT enhances early postoperative outcomes, in terms of reduction of swelling, pain relief and improvement in the function of the knee joint, compared to conventional rehabilitation without the use of KT.

DETAILED DESCRIPTION:
Kinesiotaping and Rehabilitation after Total Knee Replacement The effectiveness of Kinesiotaping (KT) in postoperative rehabilitation remains scientifically unproven, despite its widespread use. KT is believed to reduce pain and swelling, improve muscle function, and enhance joint mobility by promoting blood flow and lymphatic drainage. However, high-quality studies assessing its efficacy, particularly following Total Knee Replacement (TKR), are lacking.

Aim of the Study The aim of this study is to demonstrate that KT, when applied during inpatient rehabilitation after TKR, improves clinical outcomes compared to standard rehabilitation without KT.

Specifically, the investigators aim to show that:

KT reduces postoperative swelling and pain, thereby enhancing knee function. KT promotes faster recovery of muscle strength and range of motion. KT shortens the time needed to achieve key postoperative milestones, allowing for a more effective rehabilitation process.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Patients who have undergone primary Total Knee Replacement (TKR) with uncomplicated wound conditions.
* No signs of infection post-surgery.
* Ability to understand study procedures and complete required questionnaires.

Exclusion Criteria:

* Revision TKR surgeries.
* Early postoperative complications (e.g., wound healing disorders, deep infections, thrombosis).
* Severe comorbidities (e.g., heart failure NYHA class 3-4, renal insufficiency grade 3-4, chronic lymphedema, dermatological conditions).
* Known allergies to Kinesiotaping (KT) or adhesive materials.
* Neurological or neuromuscular disorders.
* Cognitive impairments (e.g., dementia) affecting compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain Level Using the Numeric Rating Scale (NRS) | From postoperative day 10 to postoperative day 25.
  Pain Level Using the Numeric Rating Scale (NRS): Pain intensity will be assessed using the Numeric Rating Scale, ranging from 0 (no pain) to 10 (worst possible pain).
  Unit of Measure: NRS score (0-10), where higher scores indicate worse pain.
Knee Circumference (Swelling) | From postoperative day 10 to postoperative day 25.
  Knee Circumference (Swelling): The circumference of the operated knee will be measured using a standard tape measure at a consistent anatomical location.
  Unit of Measure: Centimeters.
Passive Range of Motion (PROM) | From postoperative day 10 to postoperative day 25.
  Passive Range of Motion (PROM): Knee joint mobility (flexion and extension) will be measured using a goniometer.
  Unit of Measure: Degrees.

SECONDARY OUTCOMES:
Timed Up and Go Test | From postoperative day 10 to postoperative day 25.
  Timed Up and Go Test: Measures the time (in seconds) for a patient to rise from a chair, walk 3 meters, turn, and return to the chair.
  Unit of Measure: Seconds (lower scores indicate better mobility).
Chair Stand Test | From postoperative day 10 to postoperative day 25.
  Chair Stand Test: Measures the number of times a patient can rise from a chair and sit down within 30 seconds.
  Unit of Measure: Count (higher scores indicate better lower limb strength).
10-Meter Walk Test | From postoperative day 10 to postoperative day 25.
  10-Meter Walk Test: Measures the time taken to walk 10 meters at a self-selected pace.
  Unit of Measure: Seconds (lower scores indicate better walking ability).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Veihelmann, MD, PhD, Study Director — 1 SRH Health-center, Bad Herrenalb, Germany 2 Department of Orthopaedics, Physical Medicine & Rehabilitation, Ludwig-Maximilians- University of Munich, Munich, Germany 3 Department for Spine Therapy, Sports Hospital Stuttgart, Stuttgart, Germany
Locations (1):
- SRH Health Center Bad Herrenalb, Bad Herrenalb, Bad Herrenalb, Germany

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified individual participant data that underlie the results reported in the publication, including data on primary and secondary outcomes (e.g., pain levels, knee circumference, range of motion, functional tests). Access to data will be available upon reasonable request to researchers conducting relevant studies. Data will be shared following publication and will be accessible for up to 5 years. Researchers must submit a formal proposal, and data sharing agreements will be required to protect privacy and confidentiality.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code